CLINICAL TRIAL: NCT06258551
Title: Dynamics of Colonization and Infection by Multidrug-Resistant Pathogens in Immunocompromised and Critically Ill Patients
Acronym: DYNAMITE
Status: Recruiting | Type: Observational
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); M.D. Anderson Cancer Center (Other); Baylor College of Medicine (Other); University of Houston (Other); William Marsh Rice University (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Cesar Arias, Professor and Chief, Division of Infectious Diseases, The Methodist Hospital Research Institute
Other Study IDs: PRO00035528; 1P01AI152999-01 (NIH)
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Antimicrobial Drug Resistance; Antibiotic Resistant Infection; Clostridium Difficile; Carbapenem-Resistant Enterobacteriaceae Infection; Extended Spectrum Beta-Lactamase Producing Bacteria Infection; Vancomycin Resistant Enterococci Infection; Carbapenem Resistant Bacterial Infection; Vancomycin-Resistant Enterococcal Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensive Care Unit: Patients admitted to an intensive care unit (No interventions administered)
- Bone Marrow Transplant Unit: Patients admitted to a cancer treatment center for allogeneic stem cell transplantation (No interventions administered)

SUMMARY:
The goal of this observational study is to investigate how bacterial populations from the intestine and mouth of patients change during the hospitalization period and evaluate if some populations of specific bacteria increase or decrease the risk of acquiring an infection or becoming colonized by pathogenic bacteria. Participants will have the following samples collected during enrollment: stool samples (maximum 2x/week), blood draws (1x/week), oral swab (1x/week).

DETAILED DESCRIPTION:
The objectives of this study are to dissect the main microbial, clinical, and antimicrobial resistance determinants that impact colonization and infection by vancomycin-resistant enterococci (VRE), extended-spectrum beta-lactamase producing Enterobacterales (ESBL-E), carbapenem-resistant Enterobacterales (CRE), and Clostridium difficile; to evaluate the role of commensal microbiota in VRE, ESBL-E/CRE, and C. difficile colonization, and to define the functional aspects of keystone microbiota and mechanisms of protection against colonization/infection.

Patients will be recruited from both intensive care units (n=500) and stem cell transplant units (n=500) and will be followed until discharge from these units, or for a maximum of four weeks. In addition to stool, blood, and oral samples, enrolled patients will have clinical data collected by chart review to evaluate colonization/infection-related clinical status, microbiological laboratory information, exposure to antibiotics, and clinical outcomes. Positive clinical cultures taken during the course of hospitalization will also be collected for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Admission to an intensive care unit or stem cell transplant unit (for allogeneic stem cell transplantation) within previous 24 hours

Exclusion Criteria:

* <18 years of age
* Pregnancy
* History of inflammatory bowel disease (Crohn's disease, ulcerative colitis)
* Gastrointestinal derivation (colostomy, ileostomy, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from the intensive care units and stem cell transplant units from two major metropolitan hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Impact of Colonization on Clinical Outcomes Using DOOR Analysis | 30 days
  A desirability of outcome ranking (DOOR) algorithm will be used to analyze the impact of colonization by any target organism (CRE/ESBL-E, VRE, or C. difficile) on 30 day clinical outcomes. DOOR outcomes will be ranked as follows: 1) alive without infection, 2) alive with infection, or 3) dead.

SECONDARY OUTCOMES:
Additional Clinical Predictors of Negative Outcomes | 30 days
  Separate univariable logistic regression models will be used to evaluate associations between each individual component of the DOOR outcome (i.e., mortality and clinical infection) and the type of colonization as well as other independent predictors of mortality (e.g., neutropenia, hemodialysis, Pitt score, among others). Variables with p < 0.10 in bivariate analysis will also be included in the logistic models to assess for independent associations with outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar A Arias, MD, PhD, Msc, Principal Investigator — The Methodist Hospital Research Institute
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data generated by the DYNAMITE projects and Functional Genomics Core will be made available to the public through presentations at scientific meetings, peer-reviewed journal publications and articles, and/or direct sharing or deposit of data into publicly accessible databases. All banked bacterial specimens (both infecting and colonizing isolates) will be made available. Single bacterial whole genome sequencing data will be submitted to the Short Read Archive (SRA) at NCBI for unassembled data, as well as GenBank for assembled data.16S and shotgun metagenomic data will be submitted to the SRA following host sequence removal, and assembled 16S amplicons will be submitted to GenBank. Proteomic raw MS data will be submitted to the Proteomics Identifications (PRIDE) Archive. Metabolomics raw MS data will be submitted to the National Metabolomics Data Repository (NMDR). All custom bioinformatics pipelines, tools, and analytical scripts will be made available in a GitHub repository.
Time Frame: Proteomic and metabolomic data will be uploaded to their respective platforms prior to any manuscript submission to peer-reviewed journals and keys to the data will be provided to reviewers. Publication of the data in these repositories, as well as genomic sequencing data and bacterial specimens, will be made publicly available upon publication of results.

REFERENCES:
- [Background] Evans SR, Rubin D, Follmann D, Pennello G, Huskins WC, Powers JH, Schoenfeld D, Chuang-Stein C, Cosgrove SE, Fowler VG Jr, Lautenbach E, Chambers HF. Desirability of Outcome Ranking (DOOR) and Response Adjusted for Duration of Antibiotic Risk (RADAR). Clin Infect Dis. 2015 Sep 1;61(5):800-6. doi: 10.1093/cid/civ495. Epub 2015 Jun 25. PMID 26113652
- [Background] van Duin D, Lok JJ, Earley M, Cober E, Richter SS, Perez F, Salata RA, Kalayjian RC, Watkins RR, Doi Y, Kaye KS, Fowler VG Jr, Paterson DL, Bonomo RA, Evans S; Antibacterial Resistance Leadership Group. Colistin Versus Ceftazidime-Avibactam in the Treatment of Infections Due to Carbapenem-Resistant Enterobacteriaceae. Clin Infect Dis. 2018 Jan 6;66(2):163-171. doi: 10.1093/cid/cix783. PMID 29020404
- [Background] Taur Y, Xavier JB, Lipuma L, Ubeda C, Goldberg J, Gobourne A, Lee YJ, Dubin KA, Socci ND, Viale A, Perales MA, Jenq RR, van den Brink MR, Pamer EG. Intestinal domination and the risk of bacteremia in patients undergoing allogeneic hematopoietic stem cell transplantation. Clin Infect Dis. 2012 Oct;55(7):905-14. doi: 10.1093/cid/cis580. Epub 2012 Jun 20. PMID 22718773
- [Background] Satlin MJ, Chavda KD, Baker TM, Chen L, Shashkina E, Soave R, Small CB, Jacobs SE, Shore TB, van Besien K, Westblade LF, Schuetz AN, Fowler VG Jr, Jenkins SG, Walsh TJ, Kreiswirth BN. Colonization With Levofloxacin-resistant Extended-spectrum beta-Lactamase-producing Enterobacteriaceae and Risk of Bacteremia in Hematopoietic Stem Cell Transplant Recipients. Clin Infect Dis. 2018 Nov 13;67(11):1720-1728. doi: 10.1093/cid/ciy363. PMID 29701766
- [Background] Caballero S, Carter R, Ke X, Susac B, Leiner IM, Kim GJ, Miller L, Ling L, Manova K, Pamer EG. Distinct but Spatially Overlapping Intestinal Niches for Vancomycin-Resistant Enterococcus faecium and Carbapenem-Resistant Klebsiella pneumoniae. PLoS Pathog. 2015 Sep 3;11(9):e1005132. doi: 10.1371/journal.ppat.1005132. eCollection 2015 Sep. PMID 26334306
- [Background] Lee KH, Han SH, Yong D, Paik HC, Lee JG, Kim MS, Joo DJ, Choi JS, Kim SI, Kim YS, Park MS, Kim SY, Yoon YN, Kang S, Jeong SJ, Choi JY, Song YG, Kim JM. Acquisition of Carbapenemase-Producing Enterobacteriaceae in Solid Organ Transplantation Recipients. Transplant Proc. 2018 Dec;50(10):3748-3755. doi: 10.1016/j.transproceed.2018.01.058. PMID 30577266
- [Background] Ulrich RJ, Santhosh K, Mogle JA, Young VB, Rao K. Is Clostridium difficile infection a risk factor for subsequent bloodstream infection? Anaerobe. 2017 Dec;48:27-33. doi: 10.1016/j.anaerobe.2017.06.020. Epub 2017 Jun 29. PMID 28669864
- See also: World Health Organization Antimicrobial Resistance Fact Sheet — https://www.who.int/news-room/fact-sheets/detail/antimicrobial-resistance